CLINICAL TRIAL: NCT05872854
Title: Treatment of Mycosis Fungoides With Hypericin Ointment and Visible Light
Acronym: RW-HPN-MF-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ellen Kim, MD (Other)
Collaborators: Soligenix (Industry)
Responsible Party: Sponsor-Investigator, Ellen Kim, MD, Principal Investigator, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05622 (UPCC); RW-HPN-MF-01 (Other: Other Identifier); 851617 (Other: IRB number)
Record Dates: First submitted 2023-04-07; First posted 2023-05-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cutaneous T Cell Lymphoma; Mycosis Fungoides
Keywords: Cutaneous T Cell Lymphoma; Mycosis Fungoides
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — hypericin; Light; TNTCFP protein

STUDY DESIGN:
Intervention Model Description: The goal of this clinical trial is to assess the benefit of continuous treatment with open label synthetic hypericin ointment (HyBryte) and visible light in patients with mycosis fungoides for up to 12 months (54 weeks).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HyBryte (0.25 % Hypericin) with Visible Light (Experimental): HyBryte (0.25 % hypericin) ointment will be applied to CTCL lesions and treated with visible light 24 (±6) hours later starting at 5 J/cm^2. Drug application/light sessions will be done twice a week (at least 2 calendar days apart) for up to 54 weeks.
  Interventions: Drug: Hypericin; Other: Visible Light

INTERVENTIONS:
Drug: Hypericin — HyBryte is synthetic hypericin formulated as a 0.25% hypericin ointment
  Other Names: HyBryte; SGX301
Other: Visible Light — After application of HyBryte (0.25% hypericin ointment), participants will be placed in a light booth containing fluorescent light bulbs to activate the HyBryte.
  Other Names: Fluorescent light

SUMMARY:
The goal of this clinical trial is to assess the benefit of continuous treatment with synthetic hypericin ointment (HyBryte) and visible light in patients with mycosis fungoides for up to 12 months (54 weeks). Funding Source: FDA OOPD.

DETAILED DESCRIPTION:
This is an open label trial in which patients will have their mycosis fungoides (MF) lesions treated twice a week with HyBryte ointment that is followed, 24 hours later (±6 hours), by activation of the drug with visible light treatment. Patients will treat all of their MF lesions (where accessible to light therapy), but 3 to 5 lesions will be identified and followed as "Index Lesions" that will be evaluated using the Composite Assessment of Index Lesion Severity (CAILS) score every 6 weeks for the up to 54 weeks of therapy. Patients will be treated until resolution, dropout for adverse events, or plateau of therapeutic response occurs. Changes in the skin scoring mechanisms such as the CAILs and mSWAT will be tabulated for each patient and assessed across all patients enrolled in the trial to determine the response profile of HyBryte and visible light treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinical diagnosis of cutaneous T-cell lymphoma (CTCL, mycosis fungoides), Stage 1A, Stage 1B, or Stage 2A.

(Stage 1 is divided into stages 1A and 1B as follows: Stage 1A: Patches, papules, and/or plaques cover less than 10% of the skin surface. Stage 1B: Patches, papules, and/or plaques cover 10% or more of the skin surface. Stage 2A: Patches, papules, and/or plaques cover any amount of skin surface. Lymph nodes are abnormal, but they are not cancerous.)

* Subjects willing to follow the clinical protocol and voluntarily give their written informed consent
* Female subjects not pregnant nor nursing and willing to undergo a pregnancy test within 21 days prior to treatment initiation and agree to use a medically accepted method of birth control such as oral contraceptives (birth control pill), Barrier method (condom plus spermicide or diaphragm plus spermicide) or abstaining from intercourse while on study

Exclusion Criteria:

* History of allergy or hypersensitivity to any of the components of SGX301
* Pregnancy or mothers who are breast-feeding
* Males and females not willing to use effective contraception
* Subjects with history of sun hypersensitivity or photosensitive dermatoses (e.g., porphyria, systemic lupus erythematosus, Sjogren's, etc.).
* Subjects whose condition is spontaneously improving.
* Subjects receiving topical steroids or other topical treatments (e.g., nitrogen mustard) on lesions for CTCL within 2 weeks of enrollment
* Subjects receiving systemic steroids, psoralen UVA radiation therapy (PUVA), narrow band UVB light therapy (NB-UVB) or carmustine (BCNU) or other systemic therapies for CTCL within 3 weeks of enrollment
* Subjects who have received electron beam irradiation within 3 months of enrollment
* Subjects with a history of significant systemic immunosuppression
* Subjects taking other investigational drugs or drugs of abuse within 30 days of enrollment
* Subject with any condition that, in the judgment of the PI, is likely to interfere with participation in the study
* Subjects receiving drugs known to cause photosensitization within 2 weeks of starting SGX301 therapy unless they have not had evidence of photosensitization after receiving a stable dose of the medication for a minimum of 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Responses of Index Lesions | Baseline up to 54 weeks
  A Treatment Response is defined as a ≥50% improvement in the Composite Assessment of Index Lesion Severity (CAILS) score score at each evaluation timepoint (every 6 weeks up to 54 weeks) when compared to the CAILS score at baseline.
  The CAILS score measures: Erythema (or redness) on a scale of 0 (no redness) to 8 (very red), Scaling on a scale of 0 (no scaling) to 8 (all of the lesion is covered by a very rough surface), Plaque Elevation on a scale of 0 (no evidence of plaque above normal skin level) to 3 (plaque shows marked elevation above normal skin level) and Surface Area on a scale of 0 (no lesion/surface area is 0 cm^2) to 18 (the lesion is larger than 300 cm^2). A lower score means a better outcome.
  The overall CAILS score is calculated by adding the total score as described above for each of the 3-5 index lesions. A lower score means a better outcome.

SECONDARY OUTCOMES:
The percent of patients achieving a Complete Response of All Lesions | Baseline up to 54 weeks
  A Complete Response is defined as a Modified Severity Weighted Assessment Tool (mSWAT) score of 0 for all lesions at each evaluation timepoint (every 6 weeks up to 54 weeks). The mSWAT is based on an estimate of the percent total area of skin with lesions based on the body surface area (BSA), and the types of lesions present (patch, plaque, or tumor). A lower score means a better outcome.
The percent of patients achieving a PGA score of 3 (moderate improvement) from baseline to end of treatment. | Baseline up to 54 weeks
  The Physician Global Assessment (PGA) represents the investigator's assessment of the overall extent of improvement or worsening of the patient's cutaneous disease compared with baseline at each evaluation timepoint (every 6 weeks up to 54 weeks). This assessment is designed to consider all cutaneous lesions, including both index and non-index lesions, using a scale of 0 to 6, as described below:
  * 0 completely clear = No evidence of disease; 100% improvement
  * 1 almost clear = Very obvious improvement (≥90% to <100%); only traces of disease remain
  * 2 marked improvement = Significant improvement (≥50 to <90% clear); some evidence of disease remains
  * 3 moderate improvement = Intermediate between marked and mild (≥25% to <50%)
  * 4 slight improvement = ≥10% to <25%; significant evidence of disease remains
  * 5 no change = Disease has not changed significantly from baseline (10 to -25%)
  * 6 condition worse = Disease is worse than baseline by ≥25%
The percent of patients achieving at least 50% change in the mSWAT (overall skin score) from baseline to end of treatment. | Baseline up to 54 weeks
  A ≥50% improvement of the Modified Severity Weighted Assessment Tool (mSWAT) score at each evaluation timepoint (every 6 weeks up to 54 weeks) when compared to the mSWAT score at baseline. The mSWAT score was previously described.
The percent of patients achieving at least 50% change in VASitch from baseline to end of treatment. | Baseline up to 54 weeks
  The Visual Analog Scale for itch (VASitch) is a self-evaluation of the amount of itch that the patient has experienced on a visual scale of 0 to 10. A lower score means less itch is experienced. Patients will be asked to to assess the amount of itch they had experienced in the previous 24 hours at every light treatment visit (2 visits per week up to 54 weeks)
The change in CAILS score for each Index Lesion from baseline to end of treatment. | Baseline up to 54 weeks.
  The CAILS score was previously described.
The time needed to achieve at least a 50% change in the cumulative CAILS score of Index Lesions from baseline. | Baseline up to 54 weeks.
  The CAILS score was previously described.
The relative change in CAILS score for lesions classified as patch compared to plaque from baseline to end of treatment. | Baseline up to 54 weeks
  The CAILS score was previously described.
The time to maximal response in cumulative CAILS score. | Baseline up to 54 weeks
  These scores were previously described.
The time to maximal response in cumulative PGA score. | Baseline up to 54 weeks
  This score was previously described.
The time to maximal response in cumulative mSWAT score. | Baseline up to 54 weeks
  This score was previously described.
The time to maximal response in cumulative VASitch score. | Baseline up to 54 weeks
  This score was previously described.
Change in Skindex-29 score at Week 12, Week 24, Week 36 and Week 54 | Baseline up to 54 weeks
  The Skindex-29 is a self-administered survey to measure the effects of skin disease on patients' quality of life. Skindex-29 inquires about how often (Never, Rarely, Sometimes, Often, All the time) during the previous four weeks the patient experienced the effect described in each item. Seven items address the Symptoms domain, ten items the Emotional domain, and twelve items the Functioning domain. All responses are transformed to a linear scale of 100, varying from 0 (no effect) to 100 (effect experienced all the time). Skindex scores are reported as three scale scores, corresponding to the three domains; a scale score is the average of a patient's responses to items in a given domain.
Change in Patient Benefit Index score at Week 12, Week 24, Week 36 and Week 54 | Baseline up to 54 weeks
  The Patient Benefit Index (PBI) is a self-administered assessment of the patient-reported benefit in the treatment of their skin disease and is calculated based on the Patient Needs Questionnaire (PNQ) at baseline and Patient Needs Questionnaire (PNQ) at treatment time point. Patients with PBI ≥ 1 are considered having at least minimum patient-relevant treatment benefit.

CONTACTS AND LOCATIONS:
Locations (1):
- Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania, United States